CLINICAL TRIAL: NCT07303842
Title: Effect of a Low Advanced Glycation End Products Diet Blood Biomarkers of Patients With Type 2 Diabetes Mellitus: Randomized Controlled Trial.
Brief Title: Effect of a Low Advanced Glycation End Products Diet of Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, ANTONIO DE PADUA MANSUR, Dr, InCor Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 52932821.9.0000.0068
Record Dates: First submitted 2025-12-11; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease (CAD)
Keywords: Carboxymethyllysine; Advanced glycation end products in food; Type 2 diabetes mellitus; Coronary artery disease; Randomized clinical trial
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator)
  Interventions: Other: Control
- Intervention group (Active Comparator)
  Interventions: Other: a low-CML diet

INTERVENTIONS:
Other: a low-CML diet — Patients were instructed to boil or cook their food, and to avoid frying, grilling, and roasting. The assessment of CML content, as well as adherence to the dietary intervention, was based on the average of the 24-Hour Recalls (R24H) and was calculated based on the previous study conducted by Uribarri and collaborators, who evaluated 549 foods, with results published in 2010. The authors estimated that 1 AGE equals 1,000 KU (kilo-units). Considering that the study was conducted with an American population, certain regional foods were not found in the table; therefore, foods with similar composition were used to quantify CML.
  Arms: Intervention group
Other: Control — Patients on their usual diet
  Arms: Control group

SUMMARY:
The present study showed that a reduction of approximately 56% in CML consumption promoted a 30% reduction in this blood biomarker. This effect was associated with increased fiber intake and reduced consumption of polyunsaturated fatty acids, trans fatty acids, and cholesterol, in addition to a positive linear correlation with lipid peroxidation, body water, and dPFGAs. This represents a potential benefit, given that these factors favor insulin resistance (IR) and vascular endothelial injury, and consequently, the processes of diabetes and atherosclerosis. Thus, reducing the daily consumption of CML in the diet, combined with preparing foods at lower temperatures, constitutes a potentially protective nutritional intervention in the context of diabetes and, especially, vascular health, with a plausible impact on the prevention of cardiometabolic complications. It is worth noting that future research for analyses of total PFGAs, specific PFGAs such as pyrraline and pentosidine, and with dPFGAs, and/or studies involving a table of dietary PFGA composition with foods of Brazilian origin are necessary due to their importance in the public health context in Brazil. Furthermore, the need for long-term studies on restricting PFGA consumption is highlighted.

ELIGIBILITY:
Inclusion Criteria: Men and women, aged between 55 and 65 years, diagnosed with T2DM, CAD, and overweight or obesity were included.

-

Exclusion Criteria:

* Patients with the following diagnoses were excluded: insulin-dependent diabetes mellitus, renal insufficiency, hepatic insufficiency, eating disorders such as binge eating, depression, and/or anxiety. In addition, patients who were eutrophic, with a body mass index (BMI) were excluded. Smokers, patients who consumed alcoholic beverages, used nutritional supplements, or had a plant-based dietary pattern were also excluded. Likewise, patients who were participating in other research protocols or who did not complete and sign the informed consent form (ICF) were excluded.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of the low-CML diet on the percentage reduction of serum CML in patients with T2DM. | Right after the blood collection
  Quantification of serum CML was performed using the OxiSelectTM Nε-(carboxymethyl) lysine Competitive ELISA kit (Cell Biolabs®), following the manufacturer's instructions.

SECONDARY OUTCOMES:
To evaluate the effect of CML reduction on body composition, through anthropometric and bioimpedance measurements. | 30 minutes, during the consultation on the first evaluation day and on Day 15 afterward.
  For the anthropometric assessment, the following variables were used: weight, height, BMI, waist and abdomen circumference. BMI, waist-to-height ratio (WHtR), and abdominal circumference were assessed according to the World Health Organization (WHO). All circumferences were performed in triplicate. Determination of body composition was performed by bioelectrical impedance analysis (BIA) using the Tanita Corporation® (BC601 2018-2020, Maeno-cho Itabashi ku, Tokyo, Japan).
To evaluate the influence of reduced CML levels on the serum concentrations of glucose, insulin, triglycerides, HDL (High-Density Lipoprotein), and LDL (Low-Density Lipoprotein). | Right after the blood collection
  The dosages of glucose,, LDL, HDL, and triglycerides were performed using a colorimetric assay on an automated Alinity C analyzer (Abbott, TX, USA), utilizing specific kits.
  Insulin dosages were performed by chemiluminescence on an automated Alinity I analyzer (Abbott), utilizing specific kits.

CONTACTS AND LOCATIONS:
Locations (1):
- Servico de Prevencao, Cardiopatia na Mulher e Reabilitacao Cardiovascular, Instituto do Coracao (InCor), Hospital das Clinicas HCFMUSP,, São Paulo, São Paulo, Brazil